CLINICAL TRIAL: NCT00199836
Title: A Pilot Study of NY-ESO-1b Peptide Plus CpG 7909 and Montanide® ISA-51 in Patients With Cancer Expressing NY-ESO-1 or LAGE-1.
Brief Title: A Pilot Study of NY-ESO-1b Peptide Plus CpG 7909 and Montanide® ISA-51 in Patients With Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-007
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Cancer; Neoplasm
Keywords: cancer vaccine; NY-ESO-1b peptide; CpG 7909; Montanide® ISA-51; LAGE-1; immune response; safety
MeSH Terms: conditions — Neoplasms | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Cancer Expressing NY-ESO-1 or LAGE-1 Antigen. (Experimental): NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51 was administered to patients with cancer expressing NY-ESO-1 or LAGE-1 antigen. The injections were given subcutaneously beginning on week 1 and repeated every three weeks for 4 injections total. There was a 3 week follow-up period after the last injection. In the absence of toxicity and progressive disease (PD), a second cycle was offered to patients who received 4 vaccinations.
  Interventions: Biological: NY-ESO-1b peptide plus CpG 7909 and Montanide® ISA-51

INTERVENTIONS:
Biological: NY-ESO-1b peptide plus CpG 7909 and Montanide® ISA-51

SUMMARY:
This cancer vaccine research study involves the injection of the NY-ESO-1b peptide along with 2 other agents to help stimulate the immune system. Peptides are small fragments of protein. NY- ESO-1 peptides are normally found in the testis and the placenta. They have also been found on various types of cancer cells. The purpose is to stimulate the immune system to react against the peptides that are found on cancer cells.

DETAILED DESCRIPTION:
This is a pilot study of patients of HLA-A2 phenotype whose tumor expresses the NY-ESO-1 or LAGE-1 antigen. Patients will receive NY-ESO-1b peptide mixed with 0.5 milliliter (mL) of Montanide® ISA-51 and 1 mg of CpG 7909 given every three weeks for four doses by subcutaneous injection. There will be a three-week follow-up period after the fourth injection making the cycle 13 weeks long. In the absence of toxicity and progressive disease, a second cycle will be offered to patients who have received four vaccinations.

The primary objective is to evaluate the immune response (antibodies, CD8+ T-cells, and DTH) and safety to vaccination with NY-ESO-1b peptide mixed with CpG 7909 and Montanide® in patients with cancer expressing NY-ESO-1 or LAGE-1. The secondary objective is to document tumor responses in patients with evaluable or measurable disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic, measurable cancer or resected high risk Stage III/IV; resected Stage II, III, or IV non-small cell lung cancer or esophageal cancer who have declined, failed, or completed standard therapy; tumor expression of NY-ESO-1 or LAGE-1 antigen; HLA-A2 positive; Karnofsky performance status greater than or equal to 60%; hematology and biochemistry laboratory results within the limits normally expected for the patient population; age greater than or equal to 18.

Exclusion Criteria:

* Clinically significant heart disease; other serious illnesses; patients with serious intercurrent illness, requiring hospitalization; patients taking immunosuppressive drugs; autoimmune disease; known HIV positivity; other active malignancy within 1 year prior to entry into the study; participation in chemotherapy, radiation therapy, or any other clinical trial involving another investigational agent within 4 weeks prior to enrollment; pregnancy or breastfeeding; women of childbearing potential: refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-09-03 (Actual); Primary Completion 2005-09-05 (Actual); Study Completion 2006-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser K Altorki, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Karbach J, Gnjatic S, Bender A, Neumann A, Weidmann E, Yuan J, Ferrara CA, Hoffmann E, Old LJ, Altorki NK, Jager E. Tumor-reactive CD8+ T-cell responses after vaccination with NY-ESO-1 peptide, CpG 7909 and Montanide ISA-51: association with survival. Int J Cancer. 2010 Feb 15;126(4):909-18. doi: 10.1002/ijc.24850. PMID 19728336

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.
Started | 14
Completed | 8
Not Completed | 6
Not completed — Progressive Disease | 5
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 11
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With NY-ESO-1 Specific Humoral Immunity as Determined by an Increase in Antibody Titer From Baseline.
Description: Blood samples were obtained at baseline (prior to the first dose), prior to the second, third and fourth injection and 2 weeks after the fourth injection in both cycles 1 and 2 for the assessment of NY-ESO-1 specific antibodies by an enzyme-linked immunosorbent assay (ELISA). A positive response was a readable optical density at 280 nm.
Time Frame: up to 27 weeks
Population: All patients who received at least one dose of NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51 and had pre- and post-treatment samples taken.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.: NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51 was administered to patients with cancer expressing NY-ESO-1 or LAGE-1 antigen. The injections were given subcutaneously beginning on week 1 and repeated every three weeks for 4 injections total. There was a 3 week follow-up period after the last injection. In the absence of toxicity and PD, a second cycle was offered to patients who received 4 vaccinations.
Arm/Group | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.
Number analyzed (Participants) | 14
Participants
  Number of patients with negative titers both pre- and post-treatment | 8
  Number of patients with positive titers both pre- and post-treatment | 5
  Number of patients with negative titers at baseline and positive titers after treatment | 1

2. Primary Outcome: Number of Patients With NY-ESO-1 Specific Cellular Immunity as Measured by an Increase in NY-ESO-1b Specific CD8+ T-cells Following Treatment.
Description: Blood samples were obtained at baseline, prior to the second, third and fourth injection and 2 weeks after the fourth injection in both cycles 1 and 2 for the assessment of NY-ESO-1b specific CD8+ T-cells by ELISPOT assays.
Time Frame: up to 27 weeks
Population: All patients who received at least one dose of NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51 and had pre- and post-treatment samples taken were included in the Cycle 1 results. Cycle 2 results include all patients who received Cycle 2 treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.
Number analyzed (Participants) | 14
Participants
  Number of patients with an increase in NY-ESO-1b specific CD8+ T-cells during cycle 1 | 4
  Number of patients without an increase in NY-ESO-1b specific CD8+ T-cells during cycle 1 | 10
  Number of patients with an increase in NY-ESO-1b specific CD8+ T-cells during cycle 2: number analyzed (Participants) | 5
  Number of patients with an increase in NY-ESO-1b specific CD8+ T-cells during cycle 2 | 5

3. Primary Outcome: Number of Patients With Delayed-Type Hypersensitivity (DTH) Skin Reactions to NY-ESO-1b Peptide
Description: 10 mcg NY-ESO-1b peptide was injected intradermally at a separate site from the vaccination at baseline and after the second and fourth injection of each cycle.
  Assessment of DTH reactions as evidenced by redness and induration was performed 48 h after injection.
  The number of patients with DTH positive skin reactions was reported at each timepoint.
Time Frame: up to 25 weeks
Population: All patients who received at least one dose of NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51 and had pre- and post-treatment assessments at the given timeframes. One patient did not have post-injection DTH testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.
Number analyzed (Participants) | 14
Participants
  Baseline: Number of Patients With DTH Skin Reactions | 2
  Baseline: Number of Patients Without DTH Skin Reactions | 12
  Week 4: number analyzed (Participants) | 13
  Week 4: Number of Patients With DTH Skin Reactions | 0
  Week 4: Number of Patients Without DTH Skin Reactions | 13
  Week 10: number analyzed (Participants) | 8
  Week 10: Number of Patients With DTH Skin Reactions | 1
  Week 10: Number of Patients Without DTH Skin Reactions | 7
  Week 19: number analyzed (Participants) | 5
  Week 19: Number of Patients With DTH Skin Reactions | 3
  Week 19: Number of Patients Without DTH Skin Reactions | 2
  Week 25: number analyzed (Participants) | 5
  Week 25: Number of Patients With DTH Skin Reactions | 1
  Week 25: Number of Patients Without DTH Skin Reactions | 4

4. Primary Outcome: Safety as Measured by the Number of Patients With Dose Limiting Toxicities (DLT)
Description: DLT was defined as the following toxicities definitely, probably, or possibly related to the administration of NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51:
  * ≥ Grade 2 autoimmune phenomena
  * Asymptomatic bronchospasm or generalized urticaria
  * ≥ Grade 3 hematological and non hematological toxicities.
Time Frame: up to 28 weeks
Population: All patients who received at least one dose of NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.: NY-ESO-1b peptide, 100 μg mixed with 1mg CpG 7909 and 0.5mL of Montanide® ISA-51 was administered to patients with cancer expressing NY-ESO-1 or LAGE-1 antigen. The injections were given subcutaneously beginning on week 1 and repeated every three weeks for 4 injections total. There was a 3 week follow-up period after the last injection. In the absence of toxicity and PD, a second cycle was offered to patients who received 4 vaccinations.
Arm/Group | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.
Number analyzed (Participants) | 14
Participants | 0

5. Secondary Outcome: Number of Patients With Tumor Responses as Measured by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Computed tomography (CT) scans were performed at screening, and during weeks 13 and 28. Response was assessed using RECIST version 1.0 (Therasse et al, J Natl Cancer Inst 2000; 92:205-16). Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions (no evaluable disease); partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria. No evidence of disease (NED): no target or non-target lesions at baseline and no new lesions identified on post-baseline scans.
Time Frame: up to 28 weeks
Population: All patients who received at least one dose of NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51 and had at least one tumor response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.
Number analyzed (Participants) | 14
Participants
  Stable Disease | 3
  Complete Response | 0
  Partial Response | 0
  No Evidence of Disease | 2
  Progressive Disease | 9

ADVERSE EVENTS:
Time Frame: Up to 28 weeks.
Description: All adverse events (AEs) occurring after signed informed consent were to be documented in the source records and on the respective AE case report form (CRF), regardless of causal relationship. Toxicity was evaluated according to the National Cancer Institute CTCAE Scale (Version 3.0).
Groups:
- Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.: NY-ESO-1b peptide, 100 μg mixed with 1 mg CpG 7909 and 0.5mL of Montanide® ISA-51 was administered to patients with cancer expressing NY-ESO-1 or LAGE-1 antigen. The injections were given subcutaneously beginning on week 1 and repeated every three weeks for 4 injections total. There was a 3 week follow-up period after the last injection of peptide. In the absence of toxicity and PD, a second cycle was offered to patients who received 4 vaccinations.
Arm/Group | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen.
All-Cause Mortality (participants affected / at risk) | 2/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen. (N=14)
Angina pectoris (Cardiac disorders) | 1
Asthenia (General disorders) | 1
Brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Convulsion (Nervous system disorders) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Cancer Expressing NY-ESO-1 or LAGE-1 Antigen. (N=14)
Abdominal pain (Gastrointestinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 3
Application site eczema (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Axillary pain (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blood lactate dehydrogenase increased (Investigations) | 1
Brain edema (General disorders) | 1
Catheter placement (Surgical and medical procedures) | 1
Chills (General disorders) | 4
Depression (Psychiatric disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnea exertional (Cardiac disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 3
Flu-like symptoms (General disorders) | 4
Gamma glutamyl transferase elevated (Hepatobiliary disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal infection (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 2
Hepatomegaly (Hepatobiliary disorders) | 1
Herpes simplex (Infections and infestations) | 1
Hypertonia (Musculoskeletal and connective tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothermia (General disorders) | 2
Inflammation (General disorders) | 1
Injection site induration (General disorders) | 2
Injection site reaction (General disorders) | 4
Karnofsky scale worsened (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Pain (General disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 4
Resection of metastasis (Surgical and medical procedures) | 2
Restlessness (Psychiatric disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sleep disturbance (Psychiatric disorders) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Weight decreased (Investigations) | 1
Wheezes (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No